# Clinical Observation Of The Gynecological Iron-Deficiency Anemia Treated With Buxue Yimu Pills

Version 2 (June, 2017)

**Research Title**: Cooperative Adenomyosis Network

Research Leader: Aijun Sun

**Contact Telephone**: 010-69155638

**RESEARCH Institution**: Peking Union Medical College Hospital, Chinese

Academy of Medicine Sciences.

#### 1.RESEARCH BACKGROUND AND PURPOSES

Buxue Yimu Pills, Ferrous Sulfate each improve anemia, but they do so by different machanisms. We generally treat patients with uncomplicated Iron Deficiency Anemia with oral iron due to the ease of administration, and Ferrous Sulfate is one of the most commonly used drugs.

Buxue Yimu Pills consists of multiple chinses herbs including Angelica Sinensis, Astragalus, Donkey-Hide Gelatin, Herba Leonuri, Citrus etc., which gains widespread application in the treatment after women's abortion or operations of uterine cavity.

This study evaluates Buxue Yimu Pills, Ferrous Sulfate and the addition of Buxue Yimu Pills to Ferrous Sulfate in the treatment of Iron-Deficiency Anemia in adult women, with the object to perform clinical efficacy and safety assessment. we expect to conduct research on its metabonomics, trying to probe into the mechanism and pharmacodyamic material basis of this mysterious traditional Chinese medicine, and finally improve more access to this therapy, promote individual treatment, and control medical cost.

#### 2.RESEARCH PROCESS AND METHODS

This study was approved by the Ethnic Committee of Peking Union Medical College Hospital, Chinese Academy of Sciences. The researcher enrolled patients according to the uniform inclusion/ exclusion criteria. To each participant, medical history and certain demographic features will be recorded, general physical examination as well as gynecologic physical examination will be performed, and some outcomes measurement needs to complete. The participants will be divided randomly into 3 groups and undergo corresponding medical treatment for 1month with a follow-up later.

## 3. POSSIBLE RISKS (OR DISCOMFORT, INCONVENIENCE)

During the research, patients need to complete relevent examinations, which require to undergo blood tests on an empty stomach for twice (12-15ml for each test). Doctor-in-charge will monitor your condition changes and drug reactions in real time. Researchers do not charge any fee to any patients.

### 4. RELEVANT DETAILS CONSULTING

You have the right to consult on relevant informations. If you want to know more details about your rights and possible risks, the consulting telephone (Ethnic Committee of Peking Union Medical College Hospital) is (010)69155817.

## 5. RIGHT TO WITHDRAW FROM THESTUDY

You have the right to withdraw at any time from the study and to request that all previous data collected be deleted.

#### 6. PRIVACY POLICY

Researchers will protect your privacy.

#### 7. STATEMENT

Taking part in this study is completely voluntary. You do not have to participate if you don't want to. You may also leave the study at any time. If you leave the study before it is finished, there will be no penalty to you, and you will not lose any benefits to which you are otherwise entitled.

I understand the information printed on this form. My questions so far have been answered. I agree to take part in this study.

| Signature (Subject) | Date |
|------------------------|------|
| Signature (Researcher) | Date |